CLINICAL TRIAL: NCT02557711
Title: The Correlation Between Clinical Examination and Ultrasound Elastography Acoustic Radiation Force Impulse Findings in Hemiplegic Patients With Elbow Flexor Spasticity After Stroke
Brief Title: The Findings of Ultrasound Elastography and ARFI in Strokes Patients With Spastic Elbow Flexor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8D0951
Record Dates: First submitted 2015-09-17; First posted 2015-09-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Cerebrovascular Accident
Keywords: spasticity; stroke; ultrasound elastography; acoustic radiation force impulse
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ultrasound elastography, acoustic radiation force impulse — Two physiatrists will perform ultrasound elastography and ARFI for intra-rater and inter-rater reliability evaluation.

SUMMARY:
The aim of this study: 1. To evaluate the correlation between the clinic tools and ultrasound elastography/ ARFI imaging in stroke patients. 2. To assess the reliability of elastography/ ARFI imaging in spasticity evaluation of stroke patients.

DETAILED DESCRIPTION:
Modified Ashworth Scale (MAS) and Modified Tardieu Scale (MTS) are the most commonly used tools for spasticity assessment. But these clinic methods cannot reveal the architecture and stiffness of muscles. In recent years, ultrasound elastography and acoustic radiation force impulse (ARFI) are used in musculoskeletal disorders, including spasticity. There are no studies about the correlation between spasticity and ultrasound elastography /ARFI imaging in stroke patients. The investigators will enroll 50 stroke patients with hemiplegia and biceps brachii muscle spasticity. One physical therapist will measure MAS and MTS for spasticity of biceps brachii muscle. Two physiatrists will perform ultrasound elastography and ARFI for intra-rater and inter-rater reliability evaluation. The evaluations of B-mode ultrasound, elastography and ARFI included Heckmatt scale, biceps brachii ratio, strain ratio, dynamic sonoelastography score, color intensity, and shear wave velocity. After performing all assessments, the investigators will analyze the correlation between the clinic tools and elastography/ ARFI imaging and evaluate the reliability of elastography/ ARFI imaging in spasticity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* stroke patients with hemiplegia and biceps brachii muscle spasticity.

Exclusion Criteria:

* elbow joint contracture deformity
* combined other neuromuscular system disease
* affected upper extremity has local infection
* patient who can't follow instruction, who is restlessness and whose elbow can't meet the positioning criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: refer from physiatrists in Kaohsiung Chang Gung Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS), Modified Tardieu Scale (MTS) | patients will be evaluated within 1 month after basic history taking and consent signing

SECONDARY OUTCOMES:
the thickness of biceps brachii | patients will be evaluated within 1 month after basic history taking and signing consent
Heckmatt scale | patients will be evaluated within 1 month after finishing history taking and consent signing
strain ratio | patients will be evaluated within 1 month after finishing history taking and consent signing
Dynamic Sonoelastography Score(DS score) | patients will be evaluated within 1 month after finishing history taking and consent signing
The mean values of the intensity of red, green, and blue on histogram of bicep brachii | patients will be evaluated within 1 month after finishing history taking and consent signing
shear wave velocity within region of interest between biceps brachii and brachialis | patients will be evaluated within 1 month after finishing history taking and consent signing

CONTACTS AND LOCATIONS:
Overall Officials: Pong Ya-Ping, MD, Study Chair — Rehabilitation
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Wijck FM, Pandyan AD, Johnson GR, Barnes MP. Assessing motor deficits in neurological rehabilitation: patterns of instrument usage. Neurorehabil Neural Repair. 2001;15(1):23-30. doi: 10.1177/154596830101500104. PMID 11527276
- [Background] Ansari NN, Naghdi S, Hasson S, Mousakhani A, Nouriyan A, Omidvar Z. Inter-rater reliability of the Modified Modified Ashworth Scale as a clinical tool in measurements of post-stroke elbow flexor spasticity. NeuroRehabilitation. 2009;24(3):225-9. doi: 10.3233/NRE-2009-0472. PMID 19458429
- [Background] Kaya T, Karatepe AG, Gunaydin R, Koc A, Altundal Ercan U. Inter-rater reliability of the Modified Ashworth Scale and modified Modified Ashworth Scale in assessing poststroke elbow flexor spasticity. Int J Rehabil Res. 2011 Mar;34(1):59-64. doi: 10.1097/MRR.0b013e32833d6cdf. PMID 20671560
- [Background] Blackburn M, van Vliet P, Mockett SP. Reliability of measurements obtained with the modified Ashworth scale in the lower extremities of people with stroke. Phys Ther. 2002 Jan;82(1):25-34. doi: 10.1093/ptj/82.1.25. PMID 11784275
- [Background] Ansari NN, Naghdi S, Moammeri H, Jalaie S. Ashworth Scales are unreliable for the assessment of muscle spasticity. Physiother Theory Pract. 2006 Jun;22(3):119-25. doi: 10.1080/09593980600724188. PMID 16848350
- [Background] Ansari NN, Naghdi S, Arab TK, Jalaie S. The interrater and intrarater reliability of the Modified Ashworth Scale in the assessment of muscle spasticity: limb and muscle group effect. NeuroRehabilitation. 2008;23(3):231-7. PMID 18560139
- [Background] Mehrholz J, Wagner K, Meissner D, Grundmann K, Zange C, Koch R, Pohl M. Reliability of the Modified Tardieu Scale and the Modified Ashworth Scale in adult patients with severe brain injury: a comparison study. Clin Rehabil. 2005 Oct;19(7):751-9. doi: 10.1191/0269215505cr889oa. PMID 16250194
- [Background] Alhusaini AA, Dean CM, Crosbie J, Shepherd RB, Lewis J. Evaluation of spasticity in children with cerebral palsy using Ashworth and Tardieu Scales compared with laboratory measures. J Child Neurol. 2010 Oct;25(10):1242-7. doi: 10.1177/0883073810362266. Epub 2010 Mar 10. PMID 20223745
- [Background] Mackey AH, Walt SE, Lobb G, Stott NS. Intraobserver reliability of the modified Tardieu scale in the upper limb of children with hemiplegia. Dev Med Child Neurol. 2004 Apr;46(4):267-72. doi: 10.1017/s0012162204000428. PMID 15077704
- [Background] Pierani A, Heguy A, Fujii H, Roeder RG. Activation of octamer-containing promoters by either octamer-binding transcription factor 1 (OTF-1) or OTF-2 and requirement of an additional B-cell-specific component for optimal transcription of immunoglobulin promoters. Mol Cell Biol. 1990 Dec;10(12):6204-15. doi: 10.1128/mcb.10.12.6204-6215.1990. PMID 2123291
- [Background] Ansari NN, Naghdi S, Hasson S, Azarsa MH, Azarnia S. The Modified Tardieu Scale for the measurement of elbow flexor spasticity in adult patients with hemiplegia. Brain Inj. 2008 Dec;22(13-14):1007-12. doi: 10.1080/02699050802530557. PMID 19117179
- [Background] Pillen S, van Keimpema M, Nievelstein RA, Verrips A, van Kruijsbergen-Raijmann W, Zwarts MJ. Skeletal muscle ultrasonography: Visual versus quantitative evaluation. Ultrasound Med Biol. 2006 Sep;32(9):1315-21. doi: 10.1016/j.ultrasmedbio.2006.05.028. PMID 16965971
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Girardi P, Manca M, Gimigliano R, Smania N. Is spastic muscle echo intensity related to the response to botulinum toxin type A in patients with stroke? A cohort study. Arch Phys Med Rehabil. 2012 Jul;93(7):1253-8. doi: 10.1016/j.apmr.2012.02.005. Epub 2012 Apr 12. PMID 22502807
- [Background] Tudisco C, Bisicchia S, Stefanini M, Antonicoli M, Masala S, Simonetti G. Tendon quality in small unilateral supraspinatus tendon tears. Real-time sonoelastography correlates with clinical findings. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):393-8. doi: 10.1007/s00167-013-2551-7. Epub 2013 Jun 16. PMID 23771348
- [Background] Buck AR, Verstraete N, Li Y, Schweizer A, Snedeker JG, Buck FM. Detection of small tendon lesions by sonoelastographic visualization of strain profile differences: initial experiences. Skeletal Radiol. 2012 Sep;41(9):1073-9. doi: 10.1007/s00256-011-1349-2. Epub 2012 Jan 5. PMID 22218832
- [Background] Wu CH, Chang KV, Mio S, Chen WS, Wang TG. Sonoelastography of the plantar fascia. Radiology. 2011 May;259(2):502-7. doi: 10.1148/radiol.11101665. Epub 2011 Feb 25. PMID 21357519
- [Background] Sconfienza LM, Silvestri E, Orlandi D, Fabbro E, Ferrero G, Martini C, Sardanelli F, Cimmino MA. Real-time sonoelastography of the plantar fascia: comparison between patients with plantar fasciitis and healthy control subjects. Radiology. 2013 Apr;267(1):195-200. doi: 10.1148/radiol.12120969. Epub 2013 Jan 7. PMID 23297327
- [Background] Niitsu M, Michizaki A, Endo A, Takei H, Yanagisawa O. Muscle hardness measurement by using ultrasound elastography: a feasibility study. Acta Radiol. 2011 Feb 1;52(1):99-105. doi: 10.1258/ar.2010.100190. PMID 21498334
- [Background] Yanagisawa O, Niitsu M, Kurihara T, Fukubayashi T. Evaluation of human muscle hardness after dynamic exercise with ultrasound real-time tissue elastography: a feasibility study. Clin Radiol. 2011 Sep;66(9):815-9. doi: 10.1016/j.crad.2011.03.012. Epub 2011 May 6. PMID 21529793
- [Background] Botar-Jid C, Damian L, Dudea SM, Vasilescu D, Rednic S, Badea R. The contribution of ultrasonography and sonoelastography in assessment of myositis. Med Ultrason. 2010 Jun;12(2):120-6. PMID 21173939
- [Background] Vasilescu D, Vasilescu D, Dudea S, Botar-Jid C, Sfrangeu S, Cosma D. Sonoelastography contribution in cerebral palsy spasticity treatment assessment, preliminary report: a systematic review of the literature apropos of seven patients. Med Ultrason. 2010 Dec;12(4):306-10. PMID 21210016
- [Background] Bhatia KS, Rasalkar DD, Lee YP, Wong KT, King AD, Yuen HY, Ahuja AT. Evaluation of real-time qualitative sonoelastography of focal lesions in the parotid and submandibular glands: applications and limitations. Eur Radiol. 2010 Aug;20(8):1958-64. doi: 10.1007/s00330-010-1756-0. Epub 2010 Apr 21. PMID 20407904
- [Background] Nightingale K, Soo MS, Nightingale R, Trahey G. Acoustic radiation force impulse imaging: in vivo demonstration of clinical feasibility. Ultrasound Med Biol. 2002 Feb;28(2):227-35. doi: 10.1016/s0301-5629(01)00499-9. PMID 11937286
- [Background] Fuchs D, Hausen A, Hoefler E, Schonitzer D, Werner ER, Dierich MP, Hengster P, Reibnegger G, Schulz T, Wachter H. Activated T cells in addition to LAV/HTLV-III infection: a necessary precondition for development of AIDS. Cancer Detect Prev Suppl. 1987;1:583-7. PMID 3500785
- [Background] Goycoolea HG, Goycoolea MV, Farfan CR. Racial and familial factors in otitis media. A point prevalence study on Easter Island. Arch Otolaryngol Head Neck Surg. 1988 Feb;114(2):147-9. doi: 10.1001/archotol.1988.01860140045018. PMID 3337770
- [Background] Bai M, Du L, Gu J, Li F, Jia X. Virtual touch tissue quantification using acoustic radiation force impulse technology: initial clinical experience with solid breast masses. J Ultrasound Med. 2012 Feb;31(2):289-94. doi: 10.7863/jum.2012.31.2.289. PMID 22298873
- [Background] Friedrich-Rust M, Romenski O, Meyer G, Dauth N, Holzer K, Grunwald F, Kriener S, Herrmann E, Zeuzem S, Bojunga J. Acoustic Radiation Force Impulse-Imaging for the evaluation of the thyroid gland: a limited patient feasibility study. Ultrasonics. 2012 Jan;52(1):69-74. doi: 10.1016/j.ultras.2011.06.012. Epub 2011 Jul 7. PMID 21788057
- [Background] Kang J, Kwon H, Cho J, Oh J, Nam K, Yoon S, Kang M, Lee S, Han S. Comparative study of shear wave velocities using acoustic radiation force impulse technology in hepatocellular carcinoma: the extent of radiofrequency ablation. Gut Liver. 2012 Jul;6(3):362-7. doi: 10.5009/gnl.2012.6.3.362. Epub 2012 May 2. PMID 22844566
- [Background] Park GY, Kwon DR. Sonoelastographic evaluation of medial gastrocnemius muscles intrinsic stiffness after rehabilitation therapy with botulinum toxin a injection in spastic cerebral palsy. Arch Phys Med Rehabil. 2012 Nov;93(11):2085-9. doi: 10.1016/j.apmr.2012.06.024. Epub 2012 Jul 7. PMID 22776155